CLINICAL TRIAL: NCT02909647
Title: Three Dimensional Digital Preoperative Planning for the Osteosynthesis of Distal Radius Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tokyo Medical University (Other)
Responsible Party: Principal Investigator, Yuichi Yoshii, Associate Professor, Tokyo Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-21
Record Dates: First submitted 2016-09-14; First posted 2016-09-21 (Estimated); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Distal Radius Fracture
MeSH Terms: conditions — Wrist Fractures | interventions — Fracture Fixation, Internal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Plan group (Active Comparator): 3D preoperative planning for the distal radius fracture was performed prior to the osteosynthesis.
  Interventions: Procedure: Preoperative planning; Procedure: Osteosynthesis
- Control group (Active Comparator): Conventional preoperative planning for the distal radius fracture was performed prior to the osteosynthesis.
  Interventions: Procedure: Preoperative planning; Procedure: Osteosynthesis

INTERVENTIONS:
Procedure: Preoperative planning — preoperative planning using 3D digital planning software or conventional template
Procedure: Osteosynthesis — osteosynthesis using volar locking plate

SUMMARY:
Background: Three dimensional (3D) digital pre-operative planning software for osteosynthesis of fractures was developed. To assess the usefulness of the 3D planning, we evaluated the accuracy of the reduction shapes and selected implants in the patients with distal radius fractures.

Methods: Thirty wrists of 30 distal radius fracture patients who underwent osteosynthesis using volar locking plates were evaluated. Fifteen wrists were treated with 3D preoperative planning as the plan group. The other fifteen wrists were treated with conventional preoperative planning as the control group. Volar tilt and radial inclination were measured after operation and compared with the healthy side wrist. In addition, preoperative planning and postoperative reductions were compared by measuring the volar tilt and radial inclination of the 3D images in the plan group. The intra-class correlation coefficient (ICC) values of the radiological parameters between healthy side wrists and injured side wrists, between preoperative planning and postoperative reductions were evaluated. For the accuracy of the implant choices, the ICCs for the screw lengths between the preoperative plan and the actual choices were evaluated in the plan group.

DETAILED DESCRIPTION:
Patients and Methods The study protocol was approved by our Institutional Review Board. Thirty wrists of 30 distal radius fracture patients who underwent osteosynthesis using locking plates (19 females, 11 males; age range 23-89, mean age 59.5 years) were evaluated. Patients were excluded if they reported a previous history of traumatic injuries to the arm. The patients were divided into two groups: 15 patients in the plan group utilized our 3D digital preoperative planning software, and 15 patients in the control group utilized standard preoperative assessment on plain radiographs and CT scans. The age, sex, and fracture types were matched between groups. According to the preoperative CT scans, fractures were classified using the AO classification system.

Preoperative Planning In the plan group, 3D digital preoperative planning and a surgical simulation were performed in order to determine the reduction and the placement of the implants in addition to the plate/screw size prior to surgery. Reduction and placement of the implants were simulated using software newly-developed by the authors (Zed-Trauma, LEXI Co., Ltd. Tokyo, Japan). Planning using this software is based on digital imaging and communications in medicine (DICOM) data from CT scans. All preoperative planning group patients had pre- and post-operative CT scans in order to compare the planned and post-operative reduction shape and placement of the implant. The CT comprised contiguous sections of 1 mm thickness. The software allows the surgeons to 1) visualize the fracture displacement, 2) simulate repositioning of the fragments, 3) place the plate and screws, 4) adjust the sizes of the implants, and 5) check the shape after the reduction and implant placement by measuring anatomical shape (Figure 1 and 2). After importing the DICOM images to the software, a 3D image of the distal radius was made. Each distal radius fracture was segmented according to the main fracture fragments using the cut function. Each fragment was repositioned in accordance with fracture lines. After repositioning the fragments, the bone shape was checked three dimensionally. Reduction of the fragment was performed to regain the volar tilt and the radial inclination, and less than 2mm step-off for the intra-articular displacement referring to the healthy side wrist X ray. Simulation of the implantation of the volar locking plate used 3D templates with variable sizes of plates and screws. The Stellar II locking plate (HOYA Technosurgical, Inc., Tokyo, Japan) was used in this study. This plate system has small, medium, and large sizes for the width, and short and long sizes for the plate length. Screw lengths from 10 to 24 mm for the distal (2.4 mm diameter), and 10 to 20 mm for the proximal (2.6 mm diameter) are available. Computer aided design models of different-sized implants were installed in the software. The plate size was chosen to cover the distal fragment maximally and not exceeded the width of the distal radius. The plans were made by a single hand surgeon. After the planning, osteosynthesis was performed under general anesthesia. During the surgery, the operator performed the reduction and the placement of the plate while comparing images between the preoperative plan and fluoroscopy. The surgeons tried to reproduce the planned position of the implant by checking the distances from the margin of the implant to the margin of the radius under fluoroscopy. The screw sizes were determined by intraoperative measurement in reference to the preoperative plan. For the screw fixation, a guide block was used to insert the distal screws.

In the control group, preoperative planning was performed using conventional posterior-anterior and lateral view radiographs. Based on the X-ray image, the plate size was chosen using the conventional template. After the planning, osteosynthesis was performed under general anesthesia in the same manner as for the plan group. The surgeries were performed by several residents and fellows under supervision of a hand surgeon.

Evaluations The planned sizes of implant were compared with the actual sizes used at operation in the plan group. The screw holes were numbered from 1 to 8 for the distal (there were 7 holes in small and medium plates, and 8 holes in a large plate), and from 1 to 3 for the proximal. The screw lengths actually chosen were recorded according to the screw number.

To evaluate the accuracy of the anatomical reduction, volar tilt and radial inclination of the post-operative wrists X-ray were compared with those of the healthy side wrist in both plan and control groups. The posterior-anterior view was obtained with the elbow flexed at 90°, the ulna perpendicular to the humerus, and the forearm in the pronated position. The lateral view was obtained with the elbow flexed at 90° and adducted against the trunk. The wrists were in a neutral position with no flexion, extension, or deviation in either view. Volar tilt was measured on a lateral view. The angle between a line along the distal radial articular surface and the line perpendicular to the longitudinal axis of the radius at the joint margin was measured as volar tilt. Radial inclination was measured on a posterior-anterior view. The angle between one line connecting the radial styloid tip and the ulnar aspect of the distal radius and a second line perpendicular to the longitudinal axis of the radius was measured as radial inclination. These radiological parameters were measured by a single hand surgeon. In addition, preoperative planning and postoperative reductions were compared by measuring the volar tilt and radial inclination of the 3D images in the plan group (Figure 3). The axis of the radius was adjusted. The angle between a line from the dorsal edge to the volar edge of the radius and the line perpendicular to the longitudinal axis of the radius was measured as 3D volar tilt. The angle between a line from the radial styloid tip to the ulnar aspect of the distal radius and the line perpendicular to the longitudinal axis of the radius was measured as 3D radial inclination.

Statistical Analysis The results are expressed as mean +/- standard deviation. An intra-class correlation coefficient (ICC) was used to evaluate the accuracy of the anatomical reduction. The ICC values of the radiological parameters (volar tilt and radial inclination) between healthy side wrists and injured side wrists after the surgery were evaluated in both the plan and control groups. In addition, the ICCs of the 3D measurements between the pre-operative plan and the post-operative 3D images were evaluated in the plan group.

For the accuracy of the implant choices, the ICCs for the screw lengths between the preoperative plan and the actual choices were evaluated. According to the previous recommendation12, ICC less than 0.40 was considered poor reproducibility, between 0.40 and 0.59 was considered moderate, between 0.60 and 0.74 was considered good, and between 0.75 and 1.00 was considered excellent. The differences between preoperative plan and postoperative reductions, healthy side and injured side after surgery were analyzed using the paired t-test. P values of <0.05 were considered significant. All analyses were performed using SPSS version 13.0 (SPSS, Chicago, IL, USA).

ELIGIBILITY:
Inclusion Criteria:

* the patients who have distal radius fracture in their unilateral wrist.

Exclusion Criteria:

* the patients who reported a previous history of traumatic injuries to the arm.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-01; Primary Completion 2024-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Intraclass correlation coefficients between preoperative plan and after surgery | 1 week
  An intra-class correlation coefficient (ICC) was used to evaluate the accuracy of the anatomical reduction. The ICC values of the radiological parameters (volar tilt and radial inclination) between healthy side wrists and injured side wrists after the surgery were evaluated in both the plan and control groups. In addition, the ICCs of the 3D measurements between the pre-operative plan and the post-operative 3D images were evaluated in the plan group.

CONTACTS AND LOCATIONS:
Overall Officials: Yuichi Yoshii, Principal Investigator — Tokyo Medical University
Locations (1):
- Tokyo Medical University Ibaraki Medical Center, Ami, Ibaraki, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yoshii Y, Ogawa T, Shigi A, Oka K, Murase T, Ishii T. Three-dimensional evaluations of preoperative planning reproducibility for the osteosynthesis of distal radius fractures. J Orthop Surg Res. 2021 Feb 12;16(1):131. doi: 10.1186/s13018-021-02278-9. PMID 33579338